CLINICAL TRIAL: NCT00783588
Title: A Phase 1B Extension Trial to Allow Repeat Dosing of Autologous CLL B Cells Transduced to Express Chimeric CD154 (ISF35) in Subjects Previously Treated in MDACC Protocol 2004-0914
Brief Title: A Phase I Extension Trial of Repeated Infusions of ISF35
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Memgen, LLC (Industry)
Responsible Party: William G. Wierda, M.D., Ph.D., M.D. Anderson Cancer Center
Organization: Memgen, Inc. (Industry)
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CLL-35-102
Record Dates: First submitted 2008-10-30; First posted 2008-10-31 (Estimated); Last update posted 2008-10-31 (Estimated); Status verified 2008-10

CONDITIONS: Chronic Lymphocytic Leukemia
Keywords: Chronic lymphocytic leukemia; CLL; Leukemia; Leukemia, Lymphocytic, Chronic, B-Cell; Leukemia, B-Cell; Immune System Diseases; ISF35; Ad-ISF35; Immunotherapy; Immune therapy; Active immune therapy
MeSH Terms: conditions — Leukemia, Lymphocytic, Chronic, B-Cell; Leukemia; Leukemia, B-Cell; Immune System Diseases

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

INTERVENTIONS:
Biological: ISF35 — Subjects participating in this study will receive up to two doses of 1x10^8, 3x10^8, or 1x10^9 autologous Ad-ISF35-transduced CLL B cells, depending on the dose they received in the previous Phase I trial.
  Other Names: Ad-ISF35; AdISF35

SUMMARY:
The study is a Phase Ib extension trial that will assess the toxicity, tolerability, and safety of up to two repeated administrations of 1x10^8, 3x10^8, or 1x10^9 autologous Ad-ISF35-transduced CLL B cells given intravenously to patients with CLL who tolerated ISF35 in the prior Phase I infusion trial at M.D. Anderson.

DETAILED DESCRIPTION:
In a previous Phase I clinical trial at M.D. Anderson, patients with CLL received an intravenous infusion of autologous leukemia cells transduced ex vivo with an adenovirus encoding the wild-type murine CD154. This treatment was well tolerated and without dose-limiting toxicity. Patients each experienced acute reductions in the leukemia-cell blood count and in the size of enlarged lymph nodes and spleen.

The infusion induced changes in circulating bystander, non-infected CLL cells and both acute and long-term clinical responses. The changes in bystander CLL cells were similar to those observed in CLL cells following ligation of CD40, which included enhanced or de novo expression of CD54, CD80, and CD86, allowing the modified CLL cells to function more effectively in presenting antigens to autologous T cells. Following CD40 ligation, CLL cells are induced to express CD95 and DR5 and to undergo changes in expression of pro- and anti-apoptotic proteins, ultimately favoring apoptosis in the CLL cells.

To build upon these results, an extension to this trial will be completed in order to assess the tolerability of repeated infusions of ISF35 and to test whether additional administrations will enhance the anti-leukemic activity exhibited in the previous Phase I trial.

ELIGIBILITY:
Inclusion Criteria:

1. Subjects must have been enrolled and tolerated the single dose ISF35 in MDACC Protocol 2004-0914.
2. Subjects must have adequate Ad-ISF35 transduced CLL B cells to allow for at least one additional treatment.
3. Women of childbearing potential (not postmenopausal for at least one year or not surgically incapable of bearing children) must agree not to become pregnant for the duration of the study. Both men and women participants must agree to use contraception for the duration of the study.
4. Subjects must have Zubrod performance status of ≤ 2.
5. Subjects must have adequate hematologic, renal, hepatic, and coagulation function:

   * Adequate hematologic function:

     * Platelet count ≥ 50,000/μl; AND
     * Hemoglobin ≥ 10 g/dl (may be supported by erythropoietin or transfusion).
   * Adequate renal function:

     * Serum creatinine ≤ 1.5 times upper limit of normal; OR
     * Measured creatinine clearance ≥ 40 mL/min/1.73 m^2.
   * Adequate hepatic function:

     * Total bilirubin ≤ 2.5 times upper limit of normal; AND
     * ALT ≤ 2.5 times upper limit of normal; AND
   * Adequate coagulation tests:

     * Prothrombin time international normalized ratio (INR) ≤ 2; AND
     * Partial thromboplastin time ≤ 1.66 times upper limit of normal
6. Subjects must give written informed consent for the Phase 1B extension trial.

Exclusion Criteria:

1. Unresolved toxicity (Grade ≥ 2) from single administration of Add-ISF35 transduced autologous CLL B cells.
2. Presence of more than 55% prolymphocytes.
3. Chemotherapy (e.g., purine analogues, alkylating agents, or corticosteroids), antibody therapy, immunotherapy, radiation therapy, or participation in any investigational drug treatment within 4 weeks of enrollment into protocol or at any time during the study.
4. Ongoing toxicity from prior anti-neoplastic therapy.
5. Prior gene therapy (EXCEPT Ad-ISF35) or allogeneic stem cell transplantation.
6. Untreated autoimmune hemolytic anemia or immune thrombocytopenia.
7. Active infection requiring parenteral antibiotics.
8. HIV/HBV/HCV seropositivity.
9. Uncompensated hypothyroidism (defined as TSH greater than 4x upper limit of normal not treated with replacement hormone).

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 4 (Actual)
Dates: Start 2007-05; Primary Completion 2008-09 (Actual); Study Completion 2008-09 (Actual)

PRIMARY OUTCOMES:
Assess the toxicity, tolerability, and safety of the repeat administration of 1x10^8, 3x10^8, or 1x10^9 autologous Ad-ISF35-transduced CLL B cells in up to 9 patients with CLL who tolerated previous treatment in MDACC Protocol 2004-0914. | Duration of the trial

SECONDARY OUTCOMES:
Assess the anti-leukemia activity of the repeat administration of Ad-ISF35 transduced CLL B cells by evaluating reduction in leukemia count, reduction in adenopathy and splenomegaly, and improvement in bone marrow function. | Duration of the trial
Assess the quality of life with repeat Ad-ISF35 treatment. | Two months
Assess pharmacodynamic endpoints including induction of T cell anti-leukemia immune responses, antibody production against autologous CLL B cells, and changes in bystander leukemia cell phenotype. | Two months

CONTACTS AND LOCATIONS:
Overall Officials: William G. Wierda, M.D., Ph.D., Principal Investigator — M.D. Anderson Cancer Center
Locations (1):
- University of Texas M.D. Anderson Cancer Center, Houston, Texas, United States

REFERENCES:
- [Background] Aguilar-Santelises M, Rottenberg ME, Lewin N, Mellstedt H, Jondal M. Bcl-2, Bax and p53 expression in B-CLL in relation to in vitro survival and clinical progression. Int J Cancer. 1996 Apr 22;69(2):114-9. doi: 10.1002/(SICI)1097-0215(19960422)69:23.0.CO;2-3. PMID 8608978
- [Background] Armitage RJ, Fanslow WC, Strockbine L, Sato TA, Clifford KN, Macduff BM, Anderson DM, Gimpel SD, Davis-Smith T, Maliszewski CR, et al. Molecular and biological characterization of a murine ligand for CD40. Nature. 1992 May 7;357(6373):80-2. doi: 10.1038/357080a0. PMID 1374165
- [Background] Bacik J, Mazumdar M, Murphy BA, Fairclough DL, Eremenco S, Mariani T, Motzer RJ, Cella D. The functional assessment of cancer therapy-BRM (FACT-BRM): a new tool for the assessment of quality of life in patients treated with biologic response modifiers. Qual Life Res. 2004 Feb;13(1):137-54. doi: 10.1023/B:QURE.0000015297.91158.01. PMID 15058795
- [Background] Banchereau J, Bazan F, Blanchard D, Briere F, Galizzi JP, van Kooten C, Liu YJ, Rousset F, Saeland S. The CD40 antigen and its ligand. Annu Rev Immunol. 1994;12:881-922. doi: 10.1146/annurev.iy.12.040194.004313. PMID 7516669
- [Background] Bosch F, Ferrer A, Lopez-Guillermo A, Gine E, Bellosillo B, Villamor N, Colomer D, Cobo F, Perales M, Esteve J, Altes A, Besalduch J, Ribera JM, Montserrat E; GELCAB (Grup per l'Estudi dels Limfomes a Catalunya i Balears). Fludarabine, cyclophosphamide and mitoxantrone in the treatment of resistant or relapsed chronic lymphocytic leukaemia. Br J Haematol. 2002 Dec;119(4):976-84. doi: 10.1046/j.1365-2141.2002.03959.x. PMID 12472576
- [Background] Caligaris-Cappio F. B-chronic lymphocytic leukemia: a malignancy of anti-self B cells. Blood. 1996 Apr 1;87(7):2615-20. No abstract available. PMID 8639876
- [Background] Cantwell MJ, Sharma S, Friedmann T, Kipps TJ. Adenovirus vector infection of chronic lymphocytic leukemia B cells. Blood. 1996 Dec 15;88(12):4676-83. PMID 8977261
- [Background] Cantwell M, Hua T, Pappas J, Kipps TJ. Acquired CD40-ligand deficiency in chronic lymphocytic leukemia. Nat Med. 1997 Sep;3(9):984-9. doi: 10.1038/nm0997-984. PMID 9288724
- [Background] Castle BE, Kishimoto K, Stearns C, Brown ML, Kehry MR. Regulation of expression of the ligand for CD40 on T helper lymphocytes. J Immunol. 1993 Aug 15;151(4):1777-88. PMID 8102152
- [Background] Castro JE, Cantwell MJ, Prusak CE, Bole J, Wierda WG, Kipps TJ. long-term followup of chronic lymphocytic leukemia patients treated with CD40-ligand (CD154) gene therapy. Blood 2003; 102(11):491a (Abstract #1790).
- [Background] Cheson BD, Bennett JM, Grever M, Kay N, Keating MJ, O'Brien S, Rai KR. National Cancer Institute-sponsored Working Group guidelines for chronic lymphocytic leukemia: revised guidelines for diagnosis and treatment. Blood. 1996 Jun 15;87(12):4990-7. No abstract available. PMID 8652811
- [Background] Chu P, Deforce D, Pedersen IM, Kim Y, Kitada S, Reed JC, Kipps TJ. Latent sensitivity to Fas-mediated apoptosis after CD40 ligation may explain activity of CD154 gene therapy in chronic lymphocytic leukemia. Proc Natl Acad Sci U S A. 2002 Mar 19;99(6):3854-9. doi: 10.1073/pnas.022604399. Epub 2002 Mar 12. PMID 11891278
- [Background] Clark EA, Ledbetter JA. How B and T cells talk to each other. Nature. 1994 Feb 3;367(6462):425-8. doi: 10.1038/367425a0. PMID 8107800
- [Background] Clavio M, Miglino M, Spriano M, Pietrasanta D, Vallebella E, Celesti L, Canepa L, Pierri I, Cavaliere M, Ballerini F, Beltrami G, Rossi E, Vimercati R, Bruni R, Congiu M, Nati S, Damasio E, Santini G, Gobbi M. First line Fludarabine treatment of symptomatic chronic lymphoproliferative diseases: clinical results and molecular analysis of minimal residual disease. Eur J Haematol. 1998 Sep;61(3):197-203. doi: 10.1111/j.1600-0609.1998.tb01084.x. PMID 9753416
- [Background] Dicker F, Kater AP, Fukuda T, Kipps TJ. Fas-ligand (CD178) and TRAIL synergistically induce apoptosis of CD40-activated chronic lymphocytic leukemia B cells. Blood. 2005 Apr 15;105(8):3193-8. doi: 10.1182/blood-2003-10-3684. Epub 2004 Aug 31. PMID 15339846
- [Background] Durie FH, Foy TM, Masters SR, Laman JD, Noelle RJ. The role of CD40 in the regulation of humoral and cell-mediated immunity. Immunol Today. 1994 Sep;15(9):406-11. doi: 10.1016/0167-5699(94)90269-0. PMID 7524518
- [Background] Finn WG, Thangavelu M, Yelavarthi KK, Goolsby CL, Tallman MS, Traynor A, Peterson LC. Karyotype correlates with peripheral blood morphology and immunophenotype in chronic lymphocytic leukemia. Am J Clin Pathol. 1996 Apr;105(4):458-67. doi: 10.1093/ajcp/105.4.458. PMID 8604688
- [Background] Forstpointner R, Dreyling M, Repp R, Hermann S, Hanel A, Metzner B, Pott C, Hartmann F, Rothmann F, Rohrberg R, Bock HP, Wandt H, Unterhalt M, Hiddemann W; German Low-Grade Lymphoma Study Group. The addition of rituximab to a combination of fludarabine, cyclophosphamide, mitoxantrone (FCM) significantly increases the response rate and prolongs survival as compared with FCM alone in patients with relapsed and refractory follicular and mantle cell lymphomas: results of a prospective randomized study of the German Low-Grade Lymphoma Study Group. Blood. 2004 Nov 15;104(10):3064-71. doi: 10.1182/blood-2004-04-1323. Epub 2004 Jul 29. PMID 15284112
- [Background] Fox JP, Brandt CD, Wassermann FE, Hall CE, Spigland I, Kogon A, Elveback LR. The virus watch program: a continuing surveillance of viral infections in metropolitan New York families. VI. Observations of adenovirus infections: virus excretion patterns, antibody response, efficiency of surveillance, patterns of infections, and relation to illness. Am J Epidemiol. 1969 Jan;89(1):25-50. doi: 10.1093/oxfordjournals.aje.a120913. No abstract available. PMID 4303049
- [Background] Han T, Ezdinli EZ, Shimaoka K, Desai DV. Chlorambucil vs. combined chlorambucil-corticosteroid therapy in chronic lymphocytic leukemia. Cancer. 1973 Mar;31(3):502-8. doi: 10.1002/1097-0142(197303)31:33.0.co;2-7. No abstract available. PMID 4693581
- [Background] Hallek M, Schmitt B, Wilhelm M, Busch R, Krober A, Fostitsch HP, Sezer O, Herold M, Knauf W, Wendtner CM, Kuse R, Freund M, Franke A, Schriever F, Nerl C, Dohner H, Thiel E, Hiddemann W, Brittinger G, Emmerich B; German Chronic Lymphocytic Leukaemia Study Group. Fludarabine plus cyclophosphamide is an efficient treatment for advanced chronic lymphocytic leukaemia (CLL): results of a phase II study of the German CLL Study Group. Br J Haematol. 2001 Aug;114(2):342-8. doi: 10.1046/j.1365-2141.2001.02959.x. PMID 11529853
- [Background] Hendry L, Bowen A, Matutes E, Swansbury J, Catovsky D. Fludarabine, cyclophosphamide and mitoxantrone in relapsed or refractory chronic lymphocytic leukemia and low grade non-Hodgkin's lymphoma. Leuk Lymphoma. 2004 May;45(5):945-50. doi: 10.1080/10428190310001639489. PMID 15291353
- [Background] Hermann P, Blanchard D, de Saint-Vis B, Fossiez F, Gaillard C, Vanbervliet B, Briere F, Banchereau J, Galizzi JP. Expression of a 32-kDa ligand for the CD40 antigen on activated human T lymphocytes. Eur J Immunol. 1993 Apr;23(4):961-4. doi: 10.1002/eji.1830230430. PMID 7681403
- [Background] Holzner B, Kemmler G, Kopp M, Nguyen-Van-Tam D, Sperner-Unterweger B, Greil R. Quality of life of patients with chronic lymphocytic leukemia: results of a longitudinal investigation over 1 yr. Eur J Haematol. 2004 Jun;72(6):381-9. doi: 10.1111/j.1600-0609.2004.00233.x. PMID 15128416
- [Background] Kato K, Santana-Sahagun E, Rassenti LZ, Weisman MH, Tamura N, Kobayashi S, Hashimoto H, Kipps TJ. The soluble CD40 ligand sCD154 in systemic lupus erythematosus. J Clin Invest. 1999 Oct;104(7):947-55. doi: 10.1172/JCI7014. PMID 10510335
- [Background] Keating MJ, Kantarjian H, Talpaz M, Redman J, McCredie KB. Fludarabine therapy in chronic lymphocytic leukemia (CLL). Nouv Rev Fr Hematol (1978). 1988;30(5-6):461-6. PMID 2464794
- [Background] Keating MJ, Kantarjian H, O'Brien S, Koller C, Talpaz M, Schachner J, Childs CC, Freireich EJ, McCredie KB. Fludarabine: a new agent with marked cytoreductive activity in untreated chronic lymphocytic leukemia. J Clin Oncol. 1991 Jan;9(1):44-9. doi: 10.1200/JCO.1991.9.1.44. PMID 1702145
- [Background] Keating MJ, Flinn I, Jain V, Binet JL, Hillmen P, Byrd J, Albitar M, Brettman L, Santabarbara P, Wacker B, Rai KR. Therapeutic role of alemtuzumab (Campath-1H) in patients who have failed fludarabine: results of a large international study. Blood. 2002 May 15;99(10):3554-61. doi: 10.1182/blood.v99.10.3554. PMID 11986207
- [Background] Keating MJ, O'Brien S, Albitar M, Lerner S, Plunkett W, Giles F, Andreeff M, Cortes J, Faderl S, Thomas D, Koller C, Wierda W, Detry MA, Lynn A, Kantarjian H. Early results of a chemoimmunotherapy regimen of fludarabine, cyclophosphamide, and rituximab as initial therapy for chronic lymphocytic leukemia. J Clin Oncol. 2005 Jun 20;23(18):4079-88. doi: 10.1200/JCO.2005.12.051. Epub 2005 Mar 14. PMID 15767648
- [Background] Koduru PR, Lichtman SM, Smilari TF, Sun T, Goh JC, Karp L, Hall W, Hashimoto S, Chiorazzi N, Broome JD. Serial phenotypic, cytogenetic and molecular genetic studies in Richter's syndrome: demonstration of lymphoma development from the chronic lymphocytic leukaemia cells. Br J Haematol. 1993 Nov;85(3):613-6. doi: 10.1111/j.1365-2141.1993.tb03357.x. PMID 8136284
- [Background] Leporrier M, Chevret S, Cazin B, Boudjerra N, Feugier P, Desablens B, Rapp MJ, Jaubert J, Autrand C, Divine M, Dreyfus B, Maloum K, Travade P, Dighiero G, Binet JL, Chastang C; French Cooperative Group on Chronic Lymphocytic Leukemia. Randomized comparison of fludarabine, CAP, and ChOP in 938 previously untreated stage B and C chronic lymphocytic leukemia patients. Blood. 2001 Oct 15;98(8):2319-25. doi: 10.1182/blood.v98.8.2319. PMID 11588025
- [Background] Montserrat E, Lopez-Lorenzo JL, Manso F, Martin A, Prieto E, Arias-Sampedro J, Fernandez MN, Oyarzabal FJ, Odriozola J, Alcala A, Garcia-Conde J, Guardia R, Bosch F. Fludarabine in resistant or relapsing B-cell chronic lymphocytic leukemia: the Spanish Group experience. Leuk Lymphoma. 1996 May;21(5-6):467-72. doi: 10.3109/10428199609093445. PMID 9172812
- [Background] Montgomery C, Pocock M, Titley K, Lloyd K. Individual quality of life in patients with leukaemia and lymphoma. Psychooncology. 2002 May-Jun;11(3):239-43. doi: 10.1002/pon.557. PMID 12112484
- [Background] Noelle RJ, Roy M, Shepherd DM, Stamenkovic I, Ledbetter JA, Aruffo A. A 39-kDa protein on activated helper T cells binds CD40 and transduces the signal for cognate activation of B cells. Proc Natl Acad Sci U S A. 1992 Jul 15;89(14):6550-4. doi: 10.1073/pnas.89.14.6550. PMID 1378631
- [Background] O'Brien S, Kantarjian H, Beran M, Smith T, Koller C, Estey E, Robertson LE, Lerner S, Keating M. Results of fludarabine and prednisone therapy in 264 patients with chronic lymphocytic leukemia with multivariate analysis-derived prognostic model for response to treatment. Blood. 1993 Sep 15;82(6):1695-700. PMID 8400226
- [Background] O'Brien SM, Kantarjian HM, Cortes J, Beran M, Koller CA, Giles FJ, Lerner S, Keating M. Results of the fludarabine and cyclophosphamide combination regimen in chronic lymphocytic leukemia. J Clin Oncol. 2001 Mar 1;19(5):1414-20. doi: 10.1200/JCO.2001.19.5.1414. PMID 11230486
- [Background] Parker SL, Tong T, Bolden S, Wingo PA. Cancer statistics, 1996. CA Cancer J Clin. 1996 Jan-Feb;46(1):5-27. doi: 10.3322/canjclin.46.1.5. PMID 8548526
- [Background] Rai KR, Peterson BL, Appelbaum FR, Kolitz J, Elias L, Shepherd L, Hines J, Threatte GA, Larson RA, Cheson BD, Schiffer CA. Fludarabine compared with chlorambucil as primary therapy for chronic lymphocytic leukemia. N Engl J Med. 2000 Dec 14;343(24):1750-7. doi: 10.1056/NEJM200012143432402. PMID 11114313
- [Background] Ranheim EA, Kipps TJ. Activated T cells induce expression of B7/BB1 on normal or leukemic B cells through a CD40-dependent signal. J Exp Med. 1993 Apr 1;177(4):925-35. doi: 10.1084/jem.177.4.925. PMID 7681471
- [Background] Ranheim EA, Cantwell MJ, Kipps TJ. Expression of CD27 and its ligand, CD70, on chronic lymphocytic leukemia B cells. Blood. 1995 Jun 15;85(12):3556-65. PMID 7540066
- [Background] Ranheim EA, Kipps TJ. Tumor necrosis factor-alpha facilitates induction of CD80 (B7-1) and CD54 on human B cells by activated T cells: complex regulation by IL-4, IL-10, and CD40L. Cell Immunol. 1995 Apr 1;161(2):226-35. doi: 10.1006/cimm.1995.1031. PMID 7535196
- [Background] ROWE WP, HUEBNER RJ, GILMORE LK, PARROTT RH, WARD TG. Isolation of a cytopathogenic agent from human adenoids undergoing spontaneous degeneration in tissue culture. Proc Soc Exp Biol Med. 1953 Dec;84(3):570-3. doi: 10.3181/00379727-84-20714. No abstract available. PMID 13134217
- [Background] Roy M, Waldschmidt T, Aruffo A, Ledbetter JA, Noelle RJ. The regulation of the expression of gp39, the CD40 ligand, on normal and cloned CD4+ T cells. J Immunol. 1993 Sep 1;151(5):2497-510. PMID 8103067
- [Background] Saville W, Kipps TJ, Cantwell MJ, et al. A phase II trial of immune therapy for chronic lymphocytic leukemia. Blood. 2003; 102(11 ):437a (Abstract #1592).
- [Background] Sawitsky A, Rai KR, Glidewell O, Silver RT. Comparison of daily versus intermittent chlorambucil and prednisone therapy in the treatment of patients with chronic lymphocytic leukemia. Blood. 1977 Dec;50(6):1049-59. PMID 336116
- [Background] Shanafelt TD, Call TG. Current approach to diagnosis and management of chronic lymphocytic leukemia. Mayo Clin Proc. 2004 Mar;79(3):388-98. doi: 10.4065/79.3.388. PMID 15008611
- [Background] Tamura N, Kobayashi S, Kato K, Bando H, Haruta K, Oyanagi M, Kuriyama M, Kipps TJ, Hashimoto H. Soluble CD154 in rheumatoid arthritis: elevated plasma levels in cases with vasculitis. J Rheumatol. 2001 Dec;28(12):2583-90. PMID 11764201
- [Background] Thall PF, Simon R. A Bayesian approach to establishing sample size and monitoring criteria for phase II clinical trials. Control Clin Trials. 1994 Dec;15(6):463-81. doi: 10.1016/0197-2456(94)90004-3. PMID 7851108
- [Background] Wierda WG, Cantwell MJ, Woods SJ, Rassenti LZ, Prussak CE, Kipps TJ. CD40-ligand (CD154) gene therapy for chronic lymphocytic leukemia. Blood. 2000 Nov 1;96(9):2917-24. PMID 11049967
- [Background] Wierda W, O'Brien S, Wen S, Faderl S, Garcia-Manero G, Thomas D, Do KA, Cortes J, Koller C, Beran M, Ferrajoli A, Giles F, Lerner S, Albitar M, Kantarjian H, Keating M. Chemoimmunotherapy with fludarabine, cyclophosphamide, and rituximab for relapsed and refractory chronic lymphocytic leukemia. J Clin Oncol. 2005 Jun 20;23(18):4070-8. doi: 10.1200/JCO.2005.12.516. Epub 2005 Mar 14. PMID 15767647
- [Background] Yang Y, Wilson JM. CD40 ligand-dependent T cell activation: requirement of B7-CD28 signaling through CD40. Science. 1996 Sep 27;273(5283):1862-4. doi: 10.1126/science.273.5283.1862. PMID 8791591
- [Background] Yeh P, Perricaudet M. Advances in adenoviral vectors: from genetic engineering to their biology. FASEB J. 1997 Jul;11(8):615-23. doi: 10.1096/fasebj.11.8.9240963.
- [Result] Wierda WG, Castro JE, Aguillon R, Sampath D, Jalayer A, McMannis J, Prussak CE, Keating M, Kipps TJ. A phase I study of immune gene therapy for patients with CLL using a membrane-stable, humanized CD154. Leukemia. 2010 Nov;24(11):1893-900. doi: 10.1038/leu.2010.191. Epub 2010 Sep 30. PMID 20882050